CLINICAL TRIAL: NCT04987268
Title: Clonal Hematopoiesis of Indeterminate Potential and Residual Cardiovascular Event Tendency After Smoking Cessation
Brief Title: CHIP and Residual Cardiovascular Event Tendency After Smoking Cessation
Acronym: CHIP-RETENTION
Status: Completed | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director of cardiology, Shenyang Northern Hospital, Shenyang Northern Hospital
Other Study IDs: CHIP RETENTION V1.0
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: ACS; Clonal Hematopoiesis of Indeterminate Potential; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Clonal Hematopoiesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current-smoking: exposure: smoking
  Interventions: Genetic: clonal hematopoiesis of indeterminate potential
- Smoking-cessation: exposure: smoking cessation
  Interventions: Genetic: clonal hematopoiesis of indeterminate potential
- non-smoking: exposure: none
  Interventions: Genetic: clonal hematopoiesis of indeterminate potential

INTERVENTIONS:
Genetic: clonal hematopoiesis of indeterminate potential — Whole-exome sequencing is performed to detect the presence of clonal hematopoiesis of indeterminate potential (CHIP)

SUMMARY:
In order to identify the association between clonal hematopoiesis of indeterminate potential (CHIP) and cardiovascular risks after smoking cessation, this study intends to recruit ACS patients undergoing complete revascularization and perform whole-exome sequencing for enrolled patients to identify the prevalence of CHIP mutations. After 1-year follow-up, the relationship of presence of CHIP mutations and the occurrence of MACCEs will be explored, irrespective of smoking cessation or not. CHIP may be a potential risk factor of poor prognosis of ACS.

ELIGIBILITY:
Inclusion Criteria:

* 1. In-patients with acute coronary syndrome to undergo PCI 2. Complete revascularization during the index hospitalization 3. Written informed consent

Exclusion Criteria:

* 1. Periprocedural complications (coronary artery dissection, perforation, myocardial infarction, stroke, death) 2. Planned coronary revascularization at discharge 3. Patients with severe chronic disease (uremia, liver cirrhosis, COPD (chronic obstructive pulmonary disease) 4. Abnormal blood counts caused by hematological diseases 5. Diagnosed malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACS patients undergoing complete revascularization
Sampling Method: Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
prevalence of CHIP mutations | 24 hours
  Whole-exome sequencing is performed to detect the presence of CHIP mutations

SECONDARY OUTCOMES:
MACCE | 1 year
  MACCE includes cardiac death, non-fatal MI, non-fatal stroke, rehospitalization due to heart failure, ischemia-driven revascularization at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Study Chair — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided